CLINICAL TRIAL: NCT03467347
Title: A Randomized, Phase 1, Open-Label Study in Healthy HIV-Negative Women to Evaluate the Pharmacokinetics, Safety and Bleeding Patterns Associated With 90-Day Use of Matrix Vaginal Rings Containing 200 mg Dapivirine and 320 mg Levonorgestrel
Brief Title: PK Study of 90-Day Use of Vaginal Rings Containing Dapivirine and Levonorgestrel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Division of AIDS, US National Institute of Allergy and Infectious Diseases (Unknown); National Institute of Mental Health (NIMH) (NIH); National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MTN-044/IPM 053/CCN019; 5UM1AI068633 (NIH)
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Healthy; Contraception; Contraceptive Usage; Women
Keywords: Healthy Women; Contraception; Vaginal Ring; dapivirine; Levonorgestrel
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VR used continuously for approximately 90 days (Experimental): One silicone elastomer vaginal ring (VR) containing the active 200 mg dapivirine (DPV) and 320 mg levonorgestrel (LNG), used continuously for approximately 90 days.
  Interventions: Drug: VR: 200 mg DPV + 320 mg LNG
- VR used cyclically for approximately 90 days (Experimental): One silicone elastomer vaginal ring (VR) containing the active 200 mg dapivirine (DPV) and 320 mg levonorgestrel (LNG), used cyclically for approximately 90 days. Use the VR for 28 days, remove for 2 days.
  Interventions: Drug: VR: 200 mg DPV + 320 mg LNG

INTERVENTIONS:
Drug: VR: 200 mg DPV + 320 mg LNG — One silicone elastomer vaginal ring (VR) containing the active ingredients dapivirine (DPV) and levonorgestrel (LNG), formulated as IPM VR: 200 mg DPV + 320 mg LNG (Ring-102)

SUMMARY:
This is a Phase I single-center, two-arm, open-label, randomized study in healthy HIV-negative women to evaluate the pharmacokinetics, safety, and bleeding patterns associated with 90-day use of matrix vaginal rings containing 200 mg Dapivirine and 320 mg Levonorgestrel.

DETAILED DESCRIPTION:
This 26 week study will be conducted at one site. The site will enroll 24 subjects. Subjects will be randomized to 1 of 2 treatment regimens:

Regimen A: vaginal ring used continuously for approximately 90 days Regimen B: vaginal ring used cyclically for approximately 90 days: used for ~28 days, then removed,washed and stored for 2 days. The same ring will be used for 2 additional cycles in a similar fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Assigned female sex at birth Note: Participants who are female at birth, who now identify as male, will not be excluded so long as they are not currently or have not been on female-to-male transition therapy 90 days prior to Enrollment.
2. Age 18 through 45 years (inclusive) at Screening, verified per site SOPs
3. Able and willing to provide written informed consent to be screened for and enrolled in MTN-044/IPM 053/CCN019
4. Able and willing to provide adequate locator information, as defined in site SOPs
5. Able to communicate in spoken and written English
6. Available for all visits and able and willing to comply with all study procedural requirements
7. Willing to abstain from receptive intercourse (vaginal, oral, sex toy/vibrator/dildo and finger stimulation) and tampon use for 24 hours preceding the Enrollment Visit and clinical visits where samples are taken and for 1 week following each cervical biopsy visit
8. Not at risk for pregnancy, defined as consistently using an effective, non-hormonal method of contraception per participant report at Enrollment, and intending to continue use of an effective, non-hormonal method for the duration of study participation. Effective methods include:

   1. Non-hormonal (e.g. copper) intrauterine device (IUD) inserted at least 28 days prior to Enrollment
   2. Consistent and correct male condom use
   3. Sterilization (of participant or partner, as defined in site SOPs)
   4. Having sex exclusively with individuals assigned female sex at birth
   5. Sexually abstinent for 90 days prior to Enrollment, and intending to remain abstinent for the duration of study participation
9. In general good health as determined by the Investigator of Record (IoR)/designee at Screening and Enrollment
10. HIV-uninfected based on testing performed at Screening and Enrollment
11. Per participant report at Screening, current regular menstrual cycles of approximately 21 to 35 days in duration with no reported intermenstrual bleeding
12. Intact uterus with at least one ovary
13. Per participant report at Screening and Enrollment, states a willingness to refrain from inserting any non-study vaginal products or objects into the vagina including, but not limited to spermicides, female condoms, diaphragms, other intravaginal rings, vaginal medications, menstrual cups, cervical caps (or any other vaginally applied barrier method), vaginal douches, lubricants and moisturizers, for the 24 hours preceding the Enrollment Visit through completion of Visit 15.
14. Participants over the age of 21 (inclusive) must have documentation of a satisfactory Pap within the past 3 years prior to Enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 (Dated November 2007) to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result
15. At Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, vaginal products or vaccines after the Screening Visit through completion of Visit 15

Exclusion Criteria:

1. Body mass index greater than 40 kg/m2 at Screening
2. Pregnant at Screening or Enrollment or plans to become pregnant during the study period Note: A documented negative pregnancy test performed by study staff is required for inclusion; however, a self-reported pregnancy is adequate for exclusion from the study.
3. Diagnosed with symptomatic urinary tract infection (UTI) or reproductive tract infection (RTI) at Screening or Enrollment
4. Diagnosed with an acute STI requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines (http://www.cdc.gov/std/treatment/) at Screening or Enrollment such as gonorrhea (GC), chlamydia, trichomonas, pelvic inflammatory disease (PID), and/or syphilis Note: Genital warts requiring treatment and frequent recurrence of herpes simplex virus (HSV) are considered exclusionary; however, infrequent HSV outbreaks are not. Genital warts requiring treatment are defined as those that cause undue burden or discomfort to the participant, including bulky size, unacceptable appearance, or physical discomfort.
5. Has a clinically apparent Grade 2 or higher pelvic exam finding (observed by study staff) at Screening or Enrollment, as per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, and/or Addendum 1 (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007]) Note: Cervical bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the IoR/designee is considered expected non-menstrual bleeding and is not exclusionary.
6. Participant report and/or clinical evidence of any of the following:

   1. Known adverse reaction to any component of the study product (ever)
   2. Chronic and/or recurrent vaginal candidiasis
   3. Has a contraindication to a progestin-only contraceptive method as defined by a category 3 or 4 condition according to the CDC U.S. Medical Eligibility Criteria for Contraceptive Use, 201643
   4. Use of hormonal contraception, including hormonal IUD and implants within the 28 days prior to Enrollment
   5. Current use or planned use of CYP3A inhibitors and inducers
   6. Current use or planned use of antibiotics and/or corticosteroids that may interact with levonorgestrel
   7. Depot medroxyprogesterone acetate (DMPA) use in the 6 months prior to Enrollment or any prior use without return of regular spontaneous menstrual cycles.
   8. Non-therapeutic injection drug use in the 12 months prior to Enrollment
   9. Post-exposure prophylaxis (PEP) for HIV exposure within the 3 months prior to Enrollment
   10. Pre-exposure prophylaxis (PrEP) for HIV prevention within the 3 months prior to Enrollment
   11. Last pregnancy outcome less than 60 days prior to Enrollment
   12. Gynecologic or genital procedure (e.g., tubal ligation, dilation and curettage, piercing) 45 days or less prior to Enrollment Note: Pap test at the Screening Visit, colposcopy and cervical biopsies for evaluation of an abnormal Pap test as well as IUD insertion/removal are not exclusionary.
   13. Currently breastfeeding or planning to breastfeed during the study period
   14. Participation in any other research study involving drugs, medical devices, vaginal products or vaccines, in the 60 days prior to Enrollment
7. Has any of the following Grade 1 or higher laboratory abnormalities at Screening Visit:

   1. AST or ALT
   2. Creatinine
   3. Hemoglobin
8. Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate the interpretation of study outcome data, or otherwise interfere with achieving the study objectives including any significant uncontrolled active or chronic medical condition.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Evaluate pharmacokinetics by assessing changes in baseline of DPV and LNG concentrations in plasma. | 90 days
Evaluate pharmacokinetics by assessing changes in baseline of DPV and LNG concentrations in cervicovaginal fluid. | 90 days
Evaluate pharmacokinetics by assessing changes in baseline of DPV concentration in cervical tissue. | 90 days

SECONDARY OUTCOMES:
Incidence of Grade 2 or higher genitourinary adverse events as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected V 2.1,or Addendum 1 Female Genital Grading Table for Use in Microbicide Studies | 90 days
Incidence of Grade 3 or higher adverse events as defined by the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Magee-Women'S Res Inst and Foundation, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Friedland BA, Gundacker H, Achilles SL, Chen BA, Hoesley C, Richardson BA, Kelly CW, Piper J, Johnson S, Devlin B, Steytler J, Kleinbeck K, Dangi B, Friend C, Song M, Mensch B, van der Straten A, Jacobson C, Hendrix CW, Brown J, Blithe D, Hiller SL; MTN-030/IPM 041 and MTN-044/IPM 053/CCN019 Protocol Teams for the Microbicide Trials Network and the Contraceptive Clinical Trials Network. Acceptability of a dapivirine levonorgestrel vaginal ring in two Phase 1 trials (MTN-030/IPM 041 and MTN-044/IPM 053/CCN019): Implications for multipurpose prevention technology development. PLoS One. 2025 Jan 14;20(1):e0312957. doi: 10.1371/journal.pone.0312957. eCollection 2025. PMID 39808648